CLINICAL TRIAL: NCT02378168
Title: Late Postconditioning After Cardiac Surgery - Bridge From Surrogate Markers to Clinical Outcome
Brief Title: 6-month Follow up After Sevoflurane Postconditioning
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK ZH 2014-0040
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Heart Surgical Procedures
Keywords: postconditioning; six month follow up; cardiac event; non-cardiac event
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Retrospective Studies

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cohort of RCT (StV 5-2007; NCT00924222): Patient group with either sevoflurane or propofol sedation of the RCT (StV 5-2007; NCT00924222)
  Interventions: Other: no intervention; retrospective study

INTERVENTIONS:
Other: no intervention; retrospective study

SUMMARY:
Retrospective analysis of a 6-month follow up within a randomised controlled study in cardiac surgery with pharmacological postconditioning (sedation on intensive care unit with sevoflurane)

DETAILED DESCRIPTION:
Introduction: In a recent randomized controlled (RCT; NCT00924222) trial the investigators demonstrated in 102 patients that late post-conditioning with sevoflurane performed in the intensive care unit (ICU) reduced myocardial injury. These patients presented with lower troponin T values on the first post-operative day compared with patients undergoing propofol sedation. In order to assess possible clinical relevant long-term implications in patients enrolled in this study, the current retrospective analysis is performed focusing on cardiac and non-cardiac events during the first six months after surgery.

Methods: All patients who had successfully completed the late post-conditioning trial were included in this follow-up. Primary and secondary endpoints were the proportion of patients experiencing cardiac and non-cardiac events, respectively. Additionally, therapeutic interventions such as initiation or change of drug therapy, interventional treatment or surgery were assessed.

ELIGIBILITY:
All patients who had successfully completed the late post-conditioning trial were included in this retrospective follow-up analysis. Written and informed consent of all patients included in the first study had to be available.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had successfully completed the late postconditioning trial (NCT00924222) were included in this retrospective follow-up analysis.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
the proportion of patients with cardiac events | 6 months after cardiac surgery
  dysrhythmias, congestive heart failure and cardiac ischemic event

SECONDARY OUTCOMES:
proportion of patients experiencing non-cardiac events | 6 months after cardiac surgery
  acute or chronic pulmonary embolism, bleeding events, infections, cerebral events, acute and chronic kidney failure, defined as glomerular filtration rate below 60 ml/min

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Beck Schimmer, Prof, Principal Investigator — University Hospital Zurich, Anesthesiology
Locations (2):
- Switzerland (2):
  - University Hospital of Zurich, Zurich
  - University Hospital Zurich, Zurich